CLINICAL TRIAL: NCT04820842
Title: A Dose-Blind Extension Study With Double-blind, Placebo-Controlled, Randomized Withdrawal Period to Evaluate the Safety and Explore the Pharmacokinetics and Pharmacodynamics of TAK-994 in Adults With Narcolepsy With Cataplexy (Narcolepsy Type 1)
Brief Title: A Study of TAK-994 in Adults With Narcolepsy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: A safety signal has emerged in Phase 2 studies of TAK-994. As an immediate precautionary measure, Takeda has suspended dosing of patients and has decided to stop Phase 2 studies early.
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-994-1504; 2021-000251-39 (EudraCT Number)
Record Dates: First submitted 2021-03-26; First posted 2021-03-29 (Actual); Results first posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Narcolepsy Type 1 (NT 1)
Keywords: Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Active Drug Extension Period: TAK-994 30 mg (Experimental): TAK-994 30 mg, twice daily (BID) tablets, orally, from Day 1 (Day 57 of previous study) to Day 56 in the Active Drug Extension Period.
  Interventions: Drug: TAK-994
- Active Drug Extension Period: TAK-994 90 mg (Experimental): TAK-994 90 mg, BID, tablets, orally, from Day 1 (Day 57 of previous study) to Day 56 in the Active Drug Extension Period.
  Interventions: Drug: TAK-994
- Active Drug Extension Period: TAK-994 180 mg (Experimental): TAK-994 180 mg, BID, tablets, orally, from Day 1 (Day 57 of previous study) to Day 56 in the Active Drug Extension Period.
  Interventions: Drug: TAK-994
- Double-blind Randomized Withdrawal Period: TAK-994 30 mg (Experimental): Following the Active Drug Extension Period, participants randomized to active treatment 30 mg, BID, meeting eligibility specification and continued to receive same dose (TAK-994, 30 mg, BID, tablets, orally) from Day 57 to Day 84 in the Double-blind Randomized Withdrawal Period.
  Interventions: Drug: TAK-994
- Double-blind Randomized Withdrawal Period: TAK-994 90 mg (Experimental): Following the Active Drug Extension Period, participants randomized to active treatment 90 mg, BID, meeting eligibility specification and continued to receive same dose (TAK-994, 90 mg, BID, tablets, orally) from Day 57 to Day 84 in the Double-blind Randomized Withdrawal Period.
  Interventions: Drug: TAK-994
- Double-blind Randomized Withdrawal Period: TAK-994 180 mg (Experimental): Following the Active Drug Extension Period, participants randomized to active treatment 180 mg, BID, meeting eligibility specification and continued to receive same dose (TAK-994, 180 mg, BID, tablets, orally) from Day 57 to Day 84 in the Double-blind Randomized Withdrawal Period.
  Interventions: Drug: TAK-994
- Double-blind Randomized Withdrawal Period: Placebo (Placebo Comparator): Following the Active Drug Extension Period participants meeting eligibility specification and received placebo-matching tablets for 4 weeks (from Day 57 to Day 84) in the Double-blind Randomized Withdrawal Period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TAK-994 — TAK-994 tablets.
  Arms: Active Drug Extension Period: TAK-994 180 mg; Active Drug Extension Period: TAK-994 30 mg; Active Drug Extension Period: TAK-994 90 mg; Double-blind Randomized Withdrawal Period: TAK-994 180 mg; Double-blind Randomized Withdrawal Period: TAK-994 30 mg; Double-blind Randomized Withdrawal Period: TAK-994 90 mg
Drug: Placebo — Placebo-matching tablets.
  Arms: Double-blind Randomized Withdrawal Period: Placebo

SUMMARY:
Adults with narcolepsy who have completed the TAK-994-1501 study will be able to take part in this study.

The main aim of this study is to check if participants have side effects from TAK-994.

Participants will take one of 3 different TAK-994 dose for 8 weeks.

Then, half the participants will continue with their dose of TAK-994 and half will take a placebo. In this study, a placebo will look like a TAK-994 tablet but will not have any medicine in it. Participants will take TAK-994 or placebo for 4 weeks.

Participants will visit the clinic for a final check-up 2 weeks after their last dose of TAK-994 or placebo.

The study doctors will check for side effects from TAK-994 and placebo throughout the study.

Participants will continue to record any narcolepsy symptoms as they did in Part B of the TAK 994-1501 study.

DETAILED DESCRIPTION:
The drug being tested in the study is called TAK-994. TAK-994, is being tested to treat participants with NT1. Participants who completed Part B of TAK-994-1501(NCT04096560) will be eligible for enrollment in this study.

This study will enroll approximately 112 patients to receive one of three different TAK 994 dose for 8 weeks (active drug extension period). Participants will be randomly assigned to one of these different TAK 994 doses which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need).

Following the 8-week Active Drug Extension Period, participants will continue into a 4-week Double-blind Randomized Withdrawal Period and will receive TAK-994 or Placebo.

Participants randomized to TAK-994 will continue to receive the same dose as before.

This multi-center trial will be conducted worldwide. The duration of treatment in this study is 12 weeks plus a 2 week safety follow up period. Participants will visit the clinic 10 times after the first dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Participant with a diagnosis of Narcolepsy Type 1 (NT1) who has completed TAK-994-1501 Part B before enrollment (which will occur immediately following the final TAK-994-1501 assessments), and for whom the investigator has no clinical objection they be enrolled.

Exclusion Criteria:

1. Participant has a clinically significant moderate or severe ongoing AE related to the study drug from the prior study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2021-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (70):
- United States (35):
  - Wright Clinical Research, Alabaster, Alabama
  - Mayo Clinic Arizona 300151190, Phoenix, Arizona
  - CITrials - Bellflower, Bellflower, California
  - Santa Monica Clinical Trials, Los Angeles, California
  - Stanford School of Medicine, Redwood City, California
  - Pacific Research Network, Inc 150118105, San Diego, California
  - SDS Clinical Trials, Inc., Santa Ana, California
  - Alpine Clinical Research Center 1024762, Boulder, Colorado
  - Delta Waves Sleep Disorders and Research Center 300148510, Colorado Springs, Colorado
  - St. Francis Medical Institute, Clearwater, Florida
  - Sleep Medicine Specialists of South Florida, Miami, Florida
  - Clinical Site Partners, LLC, Miami, Florida
  - JSV Clinical Research Study, Inc, Tampa, Florida
  - Florida Pulmonary Research Institute, LLC 300127039, Winter Park, Florida
  - NeuroTrials Research, Inc. 300116336, Atlanta, Georgia
  - Sleep Practitioners, LLC Macon, Macon, Georgia
  - Clinical Research Institute 300169881, Stockbridge, Georgia
  - Hawaii Pacific Neuroscience, Honolulu, Hawaii
  - Fort Wayne Neurological Center 150711262, Fort Wayne, Indiana
  - University of Kansas Medical Center Research Institute, Inc. University of Kansas Hospital, Kansas City, Kansas
  - Helene A. Emsellem, MD PC trading as "The Center for Sleep & Wake Disorders" 150119420, Chevy Chase, Maryland
  - Beth Israel Deaconess Medical Center CardioVascular Institute, Boston, Massachusetts
  - Research Carolina Elite, Denver, North Carolina
  - Clinical Research of Gastonia, Gastonia, North Carolina
  - Raleigh Neurology Associates 300209729, Raleigh, North Carolina
  - Raleigh Neurology Associates,300209729, Raleigh, North Carolina
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Intrepid Research, Cincinnati, Ohio
  - The Cleveland Clinic Foundation 100428, Cleveland, Ohio
  - Ohio Sleep Medicine and Neuroscience Institute 186, Dublin, Ohio
  - Respiratory Specialists Berks Schuylkill Respiratory Specialists Ltd, Wyomissing, Pennsylvania
  - Medical University of South Carolina (MUSC) PARENT, Charleston, South Carolina
  - Bogan Sleep Consultants, LLC 150711087, Columbia, South Carolina
  - Sleep Therapy & Research Center 300151246, San Antonio, Texas
  - Comprehensive Sleep Medicine Associates, Sugar Land, Texas
- Canada (3):
  - West Ottawa Sleep Centre, Ottawa, Ontario
  - Toronto Sleep Institute, Toronto, Ontario
  - Jodha Tishon Inc., Toronto, Ontario
- Czechia (2):
  - Fakultni nemocnice Hradec Kralove Dept of Neurologicka klinika, Hradec Králové
  - Vseobecna fakultni nemocnice v Praze Dept of Neurologicka klinika 1.LF UK a VFN v Praze, Prague
- Finland (2):
  - Terveystalo Helsinki Uniklinikka 300186257, Helsinki
  - Turku University Hospital, Turku
- France (2):
  - Hopital Gui de Chauliac Service de Neurologie, Montpellier, Herault
  - Hopital Roger Salengro - CHU Lille service de neurologie D, Lille, Nord
- SomnoCenter Budapest, Budapest, Hungary
- Italy (4):
  - IRCCS Oasi Maria SS 300206751, Troina, Enna
  - Universita di Bologna-Clinica Neurologica-Dipartimento di Scienze Neurologiche, Bologna
  - Ospedale San Raffaele (San Raffaele Turro) Clinica Neurologica- Div Malattie del Sonno, Milan
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata U.O.C. Neurologia, Roma
- Japan (15):
  - SOUSEIKAI PS Clinic Dept of Internal Medicine, Fukuoka, Fukuoka
  - You Ariyoshi Sleep Clinic Dept of Psychiatry, Kitakyushu-shi, Fukuoka
  - Kurume University Hospital Dept of Neuropsychiatry, Kurume-shi, Fukuoka
  - Kaiseikai Kita Shin Yokohama Internal Medicine Clinic Dept of Internal Medicine, Yokohama, Kanagawa
  - Howakai Kuwamizu Hospital Dept of Internal Medicine, Kumamoto, Kumamoto
  - Jinyukai Kotorii Isahaya Hospital Dept of Psychiatry, Isahaya-shi, Nagasaki
  - Shunkaikai Inoue Hospital Dept of Respiratory Medicine, Nagasaki, Nagasaki
  - Gokeikai Osaka Kaisei Hospital Dept of Sleep Medicine, Osaka, Osaka
  - Kyowakai Hannan Hospital Dept of Psychiatry, Sakai-shi, Osaka
  - Koishikawa Tokyo Hospital Dept of Psychiatry, Bunkyō City, Tokyo-To
  - Nihon University Itabashi Hospital Dept of Neuropsychiatry, Itabashi-ku, Tokyo-To
  - Yoyogi Sleep Disorder Center Dept of Psychiatry, Shibuya-ku, Tokyo-To
  - Sleep Support Clinic Dept of Psychosomatic Medicine/Psychiatry, Shinagawa-ku, Tokyo-To
  - Sleep & Stress Clinic Dept of Psychiatry, Shinagawa-ku, Tokyo-To
  - Sumida Hospital Phase I, Sumida-ku, Tokyo-To
- South Korea (2):
  - The Catholic University of Korea, St. Vincent's Hospital 300187879, Suwon, Gyeonggi-do
  - Keimyung University Dongsan Hospital 300144594, Daegu
- Spain (4):
  - Hospital Universitario Araba Sede Santiago Sleep Unit, Vitoria-Gasteiz, Alava
  - Hospital General de Castellon Servicio de Neurofisiologia, Castellon, Castellon
  - Hospital Clinic de Barcelona Servicio de Neurologia, Barcelona
  - Hospital Vithas Nuestra Senora de America Neurofisiologia Clinica, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https:// clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/ takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Dauvilliers Y, Mignot E, Del Rio Villegas R, Du Y, Hanson E, Inoue Y, Kadali H, Koundourakis E, Meyer S, Rogers R, Scammell TE, Sheikh SI, Swick T, Szakacs Z, von Rosenstiel P, Wu J, Zeitz H, Murthy NV, Plazzi G, von Hehn C. Oral Orexin Receptor 2 Agonist in Narcolepsy Type 1. N Engl J Med. 2023 Jul 27;389(4):309-321. doi: 10.1056/NEJMoa2301940. PMID 37494485
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/60659bc6620b3b001e9dbb46

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 13 investigative sites in Spain, Italy, Japan, Korea, and the United States from 30 April 2021 to 03 November 2021 [early termination date].
Pre-assignment Details: Participants with narcolepsy type 1 (NT 1) who completed Part B of TAK-994-1501(NCT04096560) were enrolled in this study to receive TAK-994 or placebo.
Period: Active Drug Extension Period (8 Weeks)
Arm/Group | Active Drug Extension Period: TAK-994 30 mg | Active Drug Extension Period: TAK-994 90 mg | Active Drug Extension Period: TAK-994 180 mg | Double-blind Randomized Withdrawal Period: TAK-994 30 mg | Double-blind Randomized Withdrawal Period: TAK-994 90 mg | Double-blind Randomized Withdrawal Period: TAK-994 180 mg | Double-blind Randomized Withdrawal Period: Placebo
Started | 8 | 9 | 9 | 0 | 0 | 0 | 0
Completed | 5 | 1 | 2 | 0 | 0 | 0 | 0
Not Completed | 3 | 8 | 7 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor (ongoing participants in this period were discontinued) | 3 | 6 | 5 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Randomized Withdrawal Period (4 Weeks)
Arm/Group | Active Drug Extension Period: TAK-994 30 mg | Active Drug Extension Period: TAK-994 90 mg | Active Drug Extension Period: TAK-994 180 mg | Double-blind Randomized Withdrawal Period: TAK-994 30 mg | Double-blind Randomized Withdrawal Period: TAK-994 90 mg | Double-blind Randomized Withdrawal Period: TAK-994 180 mg | Double-blind Randomized Withdrawal Period: Placebo
Started | 0 | 0 | 0 | 3 | 1 | 1 | 3
Completed | 0 | 0 | 0 | 1 | 1 | 1 | 2
Not Completed | 0 | 0 | 0 | 2 | 0 | 0 | 1
Not completed — Study Terminated by Sponsor (ongoing participants in this period were discontinued) | 0 | 0 | 0 | 2 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set for the Active Drug Extension Period included all participants who were randomized and received at least 1 dose of study drug in the Active Drug Extension Period.
Groups:
- Active Drug Extension Period: TAK-994 30 mg: TAK-994 30 mg, BID tablets, orally, from Day 1 (Day 57 of previous study) to Day 56 in the Active Drug Extension Period.
- Total: Total of all reporting groups
Arm/Group | Active Drug Extension Period: TAK-994 30 mg | Active Drug Extension Period: TAK-994 90 mg | Active Drug Extension Period: TAK-994 180 mg | Total
Number analyzed (Participants) | 8 | 9 | 9 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.4 (12.13) | 31.3 (9.75) | 29.7 (11.08) | 30.8 (10.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 3 | 14
  Male | 1 | 5 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 7 | 9 | 9 | 25
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 1 | 3
  White | 6 | 6 | 6 | 18
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Spain | 4 | 1 | 0 | 5
  Italy | 1 | 4 | 4 | 9
  Japan | 1 | 0 | 1 | 2
  Korea, South | 0 | 1 | 0 | 1
  United States | 2 | 3 | 4 | 9
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 163.9 (8.39) | 170.5 (8.24) | 174.4 (6.45) | 169.8 (8.58)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 76.5 (18.52) | 81.8 (22.68) | 79.1 (16.15) | 79.2 (18.68)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per meter square (kg/m^2)] — BMI=weight (kg) / [height (m)]^2
  kilograms per meter square (kg/m^2) | 28.3 (5.86) | 27.7 (5.45) | 25.9 (5.07) | 27.3 (5.33)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One Treatment Emergent Adverse Event (TEAE) During the Active Drug Extension Period
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical investigation participants administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug whether or not it is considered related to the drug. A TEAE is defined as an AE with an onset that occurs after receiving study drug.
Time Frame: Up to 8 weeks in the Active Drug Extension Period (Weeks 1 to 8)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Active Drug Extension Period: TAK-994 30 mg | Active Drug Extension Period: TAK-994 90 mg | Active Drug Extension Period: TAK-994 180 mg
Number analyzed (Participants) | 8 | 9 | 9
Participants | 5 | 4 | 3

2. Primary Outcome: Number of Participants With at Least One Post-dose Markedly Abnormal Value (MAV) in Laboratory Test During the Active Drug Extension Period
Description: Clinical laboratory tests included hematology, serum chemistry, and urinalysis. MAV criteria: Hemoglobin <0.8×lower limit of normal (LLN), >1.2×upper limit of normal (ULN); Hematocrit <0.8×LLN, >1.2×ULN; Red blood cells (RBC) count <0.8×LLN, >1.2×ULN; White blood cells (WBC) count <0.5xLLN, >1.5xULN; Platelet count <75x10^9/liter (L), >600x10^9/L; alanine aminotransferase (ALT) >3xULN; aspartate aminotransferase (AST) >3xULN; gamma-glutamyl transferase (GGT) >3xULN; Alkaline phosphatase >3xULN; Total bilirubin >1.5xULN; Albumin <25 grams per liter (g/L); Total protein <0.8xLLN, >1.2xULN; Creatinine >1.5xULN; Blood urea nitrogen >40 milligrams per deciliters (mg/dL); Sodium <130 milliequivalents per liter (mEq/L), >150 mEq/L; Potassium <3.0 millimoles per liter (mmol/L), >5.3 mmol/L; creatine phosphokinase (CPK) >3xULN; Glucose <50 mg/dL, >300 mg/dL; Calcium <7.7 mg/dL, >11.1 mg/dL. Only categories with at least one participant with event are reported.
Time Frame: Up to 8 weeks in the Active Drug Extension Period (Weeks 1 to 8)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- Active Drug Extension Period: TAK-994 30 mg: TAK-994 30 mg, BID, tablets, orally, from Day 1 (Day 57 of previous study) to Day 56 in the Active Drug Extension Period.
Arm/Group | Active Drug Extension Period: TAK-994 30 mg | Active Drug Extension Period: TAK-994 90 mg | Active Drug Extension Period: TAK-994 180 mg
Number analyzed (Participants) | 8 | 9 | 9
Participants
  ALT: >3 x ULN | 0 | 1 | 2
  AST: >3 x ULN | 0 | 1 | 2
  Bilirubin: >1.5 x ULN | 0 | 1 | 1
  GGT: >3 x ULN | 0 | 1 | 0
  Potassium: >5.3 mmol/L | 0 | 0 | 1

3. Primary Outcome: Number of Participants With at Least One Post-dose MAV for Vital Signs During the Active Drug Extension Period
Description: MAV criteria for vital signs were: Pulse <40 beats per minute (bpm), >115 bpm; Systolic blood pressure <90 millimeters of mercury (mmHg), ≥160 mmHg; Diastolic blood pressure <50 mmHg, ≥100 mmHg, Systolic or Diastolic blood pressure change of >20, >30 mmHg from Baseline, Body temperature >38.5 degree Celsius, Respiratory Rate >21 breath/minute. Only categories with at least one participant with event are reported. Baseline for this outcome measure is Day 1 of the Active Drug Extension Period.
Time Frame: Up to 8 weeks in the Active Drug Extension Period (Weeks 1 to 8)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Active Drug Extension Period: TAK-994 30 mg | Active Drug Extension Period: TAK-994 90 mg | Active Drug Extension Period: TAK-994 180 mg
Number analyzed (Participants) | 8 | 9 | 9
Participants
  Systolic Blood Pressure: <90 mmHg | 0 | 1 | 0
  Systolic Blood Pressure: ≥160 mmHg | 0 | 1 | 0
  Systolic Blood Pressure: Change from Pre-Dose >20 mmHg | 1 | 1 | 0
  Systolic Blood Pressure: Change from Pre-Dose >30 mmHg | 0 | 1 | 0
  Diastolic Blood Pressure: ≥100 mmHg | 0 | 1 | 0
  Diastolic Blood Pressure: Change from Pre-Dose >20 mmHg | 2 | 1 | 1
  Diastolic Blood Pressure: Change from Pre-Dose >30 mmHg | 0 | 1 | 0
  Respiratory Rate: >21 breaths/minute | 1 | 0 | 2

4. Primary Outcome: Number of Participants With at Least One Post-dose MAV for Electrocardiogram (ECG) Parameters During the Active Drug Extension Period
Description: MAV criteria for ECG were: Heart rate <40 bpm, >115 bpm; PR interval ≤80 milliseconds (msec), ≥200 msec; QT interval with Fridericia correction method (QTcF) Interval ≤300 msec, >500 msec or ≥30 msec change from baseline and >450 msec; QRS duration ≤80 msec, ≥180 msec. Only categories with at least one participant with event are reported.
Time Frame: Up to 8 weeks in the Active Drug Extension Period (Weeks 1 to 8)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Active Drug Extension Period: TAK-994 30 mg | Active Drug Extension Period: TAK-994 90 mg | Active Drug Extension Period: TAK-994 180 mg
Number analyzed (Participants) | 8 | 9 | 9
Participants
  Heart Rate: <40 bpm | 1 | 0 | 1
  PR Interval: ≥200 msec | 0 | 1 | 2
  QRS Duration: ≤80 msec | 3 | 3 | 1

5. Secondary Outcome: Number of Participants With at Least One TEAE During the Double-blind Randomized Withdrawal Period
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participants administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug whether or not it is considered related to the drug. A TEAE is defined as an AE with an onset that occurs after receiving study drug.
Time Frame: Up to 4 weeks in the Double-blind Randomized Withdrawal Period (Weeks 9 to 12)
Population: Safety Analysis Set for the Double-blind Randomized Withdrawal Period included all participants who were randomized and received at least 1 dose of study drug in the Double-blind Randomized Withdrawal Period.
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Randomized Withdrawal Period: TAK-994 30 mg | Double-blind Randomized Withdrawal Period: TAK-994 90 mg | Double-blind Randomized Withdrawal Period: TAK-994 180 mg | Double-blind Randomized Withdrawal Period: Placebo
Number analyzed (Participants) | 3 | 1 | 1 | 3
Participants | 0 | 1 | 0 | 1

6. Secondary Outcome: Number of Participants With at Least One Post-dose MAV in Laboratory Test During the Double-blind Randomized Withdrawal Period
Description: Clinical laboratory tests included hematology, serum chemistry, and urinalysis. MAV criteria: Hemoglobin <0.8×LLN, >1.2×ULN; Hematocrit <0.8×LLN, >1.2×ULN; RBC count <0.8×LLN, >1.2×ULN; WBC count <0.5xLLN, >1.5xULN; Platelet count <75x10^9/L, >600x10^9/L; ALT >3xULN; AST >3xULN; GGT >3xULN; Alkaline phosphatase >3xULN; Total bilirubin >1.5xULN; Albumin <25 g/L; Total protein <0.8x LLN, >1.2xULN; Creatinine >1.5xULN; Blood urea nitrogen >40 mg/dL; Sodium <130 mEq/L, >150 mEq/L; Potassium <3.0 mmol/L, >5.3 mmol/L; CPK >3xULN; Glucose <50 mg/dL, >300 mg/dL; Calcium <7.7 mg/dL, >11.1 mg/dL.
Time Frame: Up to 4 weeks in the Double-blind Randomized Withdrawal Period (Weeks 9 to 12)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Randomized Withdrawal Period: TAK-994 30 mg | Double-blind Randomized Withdrawal Period: TAK-994 90 mg | Double-blind Randomized Withdrawal Period: TAK-994 180 mg | Double-blind Randomized Withdrawal Period: Placebo
Number analyzed (Participants) | 3 | 1 | 1 | 3
Participants | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With at Least One Post-dose MAV for Vital Signs During the Double-blind Randomized Withdrawal Period
Description: MAV criteria for vital signs were: Pulse <40 bpm, >115 bpm; Systolic blood pressure <90 mmHg, ≥160 mmHg; Diastolic blood pressure <50 mmHg, ≥100 mmHg, Systolic or Diastolic blood pressure change of >20, >30 mmHg from Baseline, Body temperature >38.5 degree Celsius, Respiratory Rate >21 breath/minute. Only categories with at least one participant with event are reported. Baseline for this outcome measure is Day 1 of the Double-blind Randomized Withdrawal Period (Day 57 of this study).
Time Frame: Up to 4 weeks in the Double-blind Randomized Withdrawal Period (Weeks 9 to 12)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Randomized Withdrawal Period: TAK-994 30 mg | Double-blind Randomized Withdrawal Period: TAK-994 90 mg | Double-blind Randomized Withdrawal Period: TAK-994 180 mg | Double-blind Randomized Withdrawal Period: Placebo
Number analyzed (Participants) | 3 | 1 | 1 | 3
Participants
  Systolic Blood Pressure: <90 mmHg | 0 | 0 | 0 | 1
  Systolic Blood Pressure: Change from Baseline >20 mmHg | 1 | 0 | 0 | 0
  Diastolic Blood Pressure: Change from Baseline >20 mmHg | 1 | 1 | 0 | 1

8. Secondary Outcome: Number of Participants With at Least One Post-dose MAV for ECG Parameters During the Double-blind Randomized Withdrawal Period
Description: MAV criteria for ECG were: Heart rate <40 bpm, >115 bpm; PR interval ≤80 msec, ≥200 msec; QTcF Interval ≤300 msec, >500 msec or ≥30 msec change from baseline and >450 msec; QRS duration ≤80 msec, ≥180 msec. Only categories with at least one participant with event are reported.
Time Frame: Up to 4 weeks in the Double-blind Randomized Withdrawal Period (Weeks 9 to 12)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Double-blind Randomized Withdrawal Period: TAK-994 30 mg | Double-blind Randomized Withdrawal Period: TAK-994 90 mg | Double-blind Randomized Withdrawal Period: TAK-994 180 mg | Double-blind Randomized Withdrawal Period: Placebo
Number analyzed (Participants) | 3 | 1 | 1 | 3
Participants | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: From randomization up to two weeks post end of treatment (up to Week 14)
Description: Safety Analysis Set for the Active Drug Extension Period and Double-blind Randomized Withdrawal Period included all participants who were randomized and received at least 1 dose of study drug in the Active Drug Extension Period and Double-blind Randomized Withdrawal Period respectively.
Groups:
- Period 1: TAK-994 30 mg BID: TAK-994 30 mg, BID tablets, orally, from Day 1 (Day 57 of previous study) to Day 56 in the Active Drug Extension Period.
- Period 1: TAK-994 90 mg BID: TAK-994 90 mg, BID, tablets, orally, from Day 1 (Day 57 of previous study) to Day 56 in the Active Drug Extension Period.
- Period 1: TAK-994 180 mg BID: TAK-994 180 mg, BID, tablets, orally, from Day 1 (Day 57 of previous study) to Day 56 in the Active Drug Extension Period.
- Period 2: TAK-994 30 mg BID: Following the Active Drug Extension Period, participants randomized to active treatment 30 mg, BID, meeting eligibility specification and continued to receive same dose (TAK-994, 30 mg, BID, tablets, orally) from Day 57 to Day 84 in the Double-blind Randomized Withdrawal Period.
- Period 2: TAK-994 90 mg BID: Following the Active Drug Extension Period, participants randomized to active treatment 90 mg, BID, meeting eligibility specification and continued to receive same dose (TAK-994, 90 mg, BID, tablets, orally) from Day 57 to Day 84 in the Double-blind Randomized Withdrawal Period.
- Period 2: TAK-994 180 mg BID: Following the Active Drug Extension Period, participants randomized to active treatment 180 mg, BID, meeting eligibility specification and continued to receive same dose (TAK-994, 180 mg, BID, tablets, orally) from Day 57 to Day 84 in the Double-blind Randomized Withdrawal Period.
- Period 2: Placebo: Following the Active Drug Extension Period participants meeting eligibility specification and received placebo-matching tablets for 4 weeks (from Day 57 to Day 84) in the Double-blind Randomized Withdrawal Period.
Arm/Group | Period 1: TAK-994 30 mg BID | Period 1: TAK-994 90 mg BID | Period 1: TAK-994 180 mg BID | Period 2: TAK-994 30 mg BID | Period 2: TAK-994 90 mg BID | Period 2: TAK-994 180 mg BID | Period 2: Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/9 | 0/9 | 0/3 | 0/1 | 0/1 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/8 | 1/9 | 1/9 | 0/3 | 0/1 | 0/1 | 0/3
Other Adverse Events (participants affected / at risk) | 5/8 | 4/9 | 3/9 | 0/3 | 1/1 | 0/1 | 1/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1: TAK-994 30 mg BID (N=8) | Period 1: TAK-994 90 mg BID (N=9) | Period 1: TAK-994 180 mg BID (N=9) | Period 2: TAK-994 30 mg BID (N=3) | Period 2: TAK-994 90 mg BID (N=1) | Period 2: TAK-994 180 mg BID (N=1) | Period 2: Placebo (N=3)
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1: TAK-994 30 mg BID (N=8) | Period 1: TAK-994 90 mg BID (N=9) | Period 1: TAK-994 180 mg BID (N=9) | Period 2: TAK-994 30 mg BID (N=3) | Period 2: TAK-994 90 mg BID (N=1) | Period 2: TAK-994 180 mg BID (N=1) | Period 2: Placebo (N=3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nervousness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Temperature intolerance (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2021-02-03): https://cdn.clinicaltrials.gov/large-docs/42/NCT04820842/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-25): https://cdn.clinicaltrials.gov/large-docs/42/NCT04820842/SAP_001.pdf